CLINICAL TRIAL: NCT06137625
Title: Rhythm Effect on Dance Learning and Associated Functions in Typical Development Children and Children With Motor Disorders.
Brief Title: Rhythm Effect on Dance Learning in Typical Development Children and Children With Motor Disorders.
Acronym: DANS-APP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RC31/22/0039; ANR-21-CE28-0031 (Other Grant/Funding Number: Agence Nationale de la Recherche (ANR))
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor disorders (Experimental): Children with motor disporders
  Interventions: Behavioral: With regular rhythm; Behavioral: Without regular rhythm
- Typical developing (Active Comparator): Typical developing children
  Interventions: Behavioral: With regular rhythm; Behavioral: Without regular rhythm

INTERVENTIONS:
Behavioral: With regular rhythm — All children learn one dance choreographie with regular rhythm music.The pre-recorded choreography is displayed on a large screen in front of the child. The child practices the choreography by imitating the models in order to learn the sequence movements.
Behavioral: Without regular rhythm — All children learn one dance choreographie without regular rhythm music.The pre-recorded choreography is displayed on a large screen in front of the child. The child practices the choreography by imitating the models in order to learn the sequence movements.

SUMMARY:
Cerebral Palsy (CP) or Developmental Coordination Disorder (DCD) leads to motor troubles impacting the everyday life, social participation and academic difficulty . According to some authors, CP and DCD pertain to a same continuum of motor disorders (MD) (Pearsall-Jones et al., 2010).Those children show an alteration in Perceptivo-Motor Procedural Learning (PMPL), corresponding to the acquisition of everyday life skill (for CP: Gagliardi et al., 2011; Gofer-Levi et al., 2013; for DCD: Gheysen et al., 2011; Blais et al., 2018). Also, recommended rehabilitation for this population are based on procedural learnings (for CP: Novak et al., 2013; for DCD: Blank et al., 2019; Inserm, 2019). It's true for dancing which present high evidence to enhance motor, cognitive, psychoaffective and social functions of this children (Cherriere, Martel, et al., 2020; Cherriere, Robert, et al., 2020). Dance is a physical activity that involve procedural learning to memorise movement sequences (choreography). Rhythm can be define as a stimuli repetition at a regular interval (Grahn & Brett, 2007; Patel, 2003). Recently studies tend to shown that rhythm is essential to enhance motor control and procedural learning (Ghai et al., 2022; Lagarrigue et al., 2021). To validate this hypothesis, the investigators will evaluate typical development children and children with CP MD learning of a dance choreography with and without rhythm.

ELIGIBILITY:
Inclusion Criteria:

For all the participants:

* Aged from 8 to 16 include.
* Free, informed, written, and signed consent of the holders of parental authority
* Free and informed consent of the minor
* Affiliation with or benefiting from a social security scheme.
* Ability to understand the instructions (investigator's assessment)

For the participant with Motor disorders (MD):

1. For children with CP:

   * CP diagnosis
   * Gross Motor Function Classification System level between I to IV.
   * Manual Ability Classification System level between I to IV.
2. For children with DCD:

   * A diagnosis of DCD

For the participant with typical development:

* No CP diagnosis
* No neurological trouble nor functional disfunction including developmental coordination disorder.

Exclusion Criteria:

* -Autism spectrum disorder diagnosed according to the DSM-5 (APA, 2015)
* Hearing deficiency diagnosed according to the DSM-5 (APA, 2015) or uncorrected hearing deficiency that doesn't allows the participant to hear a music with a sound level between 45 and 70 decibels.
* Visual deficiency diagnosed according to the DSM-5 (APA, 2015)
* Intellectual developmental disorder diagnosed according to the DSM-5 (APA, 2015)
* Behavioural disorders diagnosed according to the DSM-5 (APA, 2015)
* Diagnosed epilepsia
* Pregnancy (check in young pubescent and sexually active women) or breastfeeding.
* Children already include in ongoing interventional study.
* Children with both parent who benefit of legal protection (guardianship, curatorship, safeguard of justice).

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Retention score of the choreography | Day 0
  Number of movements in the choreography performed correctly and in order after practice is analysed by video using a standardised observation grid scored independently and blind to the condition by two trained judges.

SECONDARY OUTCOMES:
the effect of regular rhythm on Perceptivo-Motor Procedural Learning (PMPL) | Day 0
  The PMPL is measured by an informatised and standardised test (EVAL_App_Kids test)
the effect of regular rhythm on sensorimotor function | Day 0
  the effect is measured by rhythm perception and production task
the effect of regular rhythm on cognitive function | Day 0
  the effect is measured by informatised test on attention and executive function
the effect of regular rhythm on psychoaffective function | Day 0
  the effect is measured by Intrinsic Motivation Inventory questionnaire (IMI)

CONTACTS AND LOCATIONS:
Locations (1):
- Toulouse Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No